CLINICAL TRIAL: NCT05118126
Title: Diagnostic and Therapeutic Value of Gut Microbiome in Adult Immune Thrombocytopenia
Brief Title: Gut Microbiota in ITP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University People's Hospital (Other)
Collaborators: Beijing Hospital (Other Government)
Responsible Party: Principal Investigator, Xiao Hui Zhang, Vice president of Peking Univeristy Institute of Hematology, Peking University People's Hospital
Other Study IDs: PKU-ITP033
Record Dates: First submitted 2021-11-01; First posted 2021-11-11 (Actual); Last update posted 2022-01-12 (Actual); Status verified 2022-01

CONDITIONS: ITP

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Fecal sample collection and metagenomic sequencing: A specific stool sample collector was selected to collect an appropriate amount of stool samples (≥1g/ sample). Samples that could not be extracted immediately were transported on dry ice and stored at -80℃. DNA was extracted by phenol/chloroform method. Qubit Fluorometer is used to test samples DNA concentration, agarose gel electrophoresis (gel concentration: 1%; Voltage: 150 V; Electrophoresis time: 40 min) is used to test DNA integrity of samples, and unqualified samples with insufficient DNA amount or degradation were eliminated. Qualified samples were used for DNA library construction and Illumina sequencing. The sequencing library was constructed according to Illumina's official operating instructions and further optimized. Qualified libraries were sequenced using Illumina platform.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Prospective, observational study to explore the significance of gut microbiome in the diagnosis of ITP, and to identify the predictive value of baseline gut microbiome for GC resistance/relapse.

DETAILED DESCRIPTION:
A prospective, observational study to (1) collect fecal samples from ITP patients at initial diagnosis (baseline) and after first-line GC treatment, (2) detect the composition of gut microbiome and related metabolites using metagenomic sequencing combined with metabolomics, (3) observe the impact of first-line treatment on gut microbiome, (4) explore the significance of gut microbiome in the diagnosis of ITP, and (5) identify the predictive value of baseline gut microbiome for GC resistance/relapse, thus to provide new ideas for clinical diagnosis and treatment of ITP.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older;
* Isolated thrombocytopenia (platelet count of less than 100×10^9/L);
* Normal leukocyte and erythrocyte counts according to routine blood tests;
* Did not receive any medication for thrombocytopenia for 6 months.

Exclusion Criteria:

* Secondary ITP such as drug-associated thrombocytopenia;
* Thrombocytopenia caused by viral infection (HIV, Hepatitis B virus or Hepatitis C virus);
* Nursing or pregnant women;
* Severe dysfunction of the heart, kidney, lung or liver;
* Active or previous malignancy;
* Patients with other diseases were undergoing treatment with immunosuppressants;
* Myelodysplastic disorder or myelofibrosis;
* Patients who were undergoing first - or second-line therapy for thrombocytopenia within 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with newly diagnosed ITP who would receive first-line therapy (glucocorticoid therapy with platelet infusion) according to the clinician's or patient's decision.
Sampling Method: Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2022-01 (Estimated); Primary Completion 2022-06 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
AUC value of 1-month drug resistance/relapse using baseline gut microbiota efficacy prediction model | 1 month
  The prediction model is constructed and calculated using machine learning methods

SECONDARY OUTCOMES:
AUC value of 3-month drug resistance/relapse using baseline gut microbiota efficacy prediction model | 3 months
  The prediction model is constructed and calculated using machine learning
AUC value of 6-month drug resistance/relapse using baseline gut microbiota | 6 months
  The prediction model is constructed and calculated using machine learning
Time to response | 6 months
  The time to achieve platelet count ≥ 30×10^9/L and at least 2-fold increase of the baseline count and absence of bleeding since start of treatment.
Duration of response | 6 months
  The duration of achieve platelet count ≥ 30×10^9/L and at least 2-fold increase of the baseline count and absence of bleeding since start of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Xiao-Hui Zhang, Dr., Principal Investigator — Peking University People's Hospital, Peking University Insititute of Hematology
Locations (1):
- Peking University Insititute of Hematology, Peking University People's Hospital, Beijing, Beijing Municipality, China